CLINICAL TRIAL: NCT06529614
Title: A New Detection Method for MicroRNA in Patients With Breast Cancer
Brief Title: An In-situ Detection for MicroRNA
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lei Dou, Dr., Tongji Hospital
Other Study IDs: 20240771
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Health donor group
  Interventions: Other: In-situ detection for Micro-RNA
- Breast cancer group
  Interventions: Other: In-situ detection for Micro-RNA

INTERVENTIONS:
Other: In-situ detection for Micro-RNA — a new in-situ detection methods for Micro-RNA

SUMMARY:
We designed a new in-site detection method for MicroRNA in the serum of patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria: Healthy without serious diseases

-

Exclusion Criteria:

* situations that may affect the results

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who have diagnosed with breat cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of test | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Shabei Xu, Dr., Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No